CLINICAL TRIAL: NCT02572076
Title: Clinical Investigational Plan: Evaluation of the Performance of the Motus Cleansing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL00035
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2016-12

CONDITIONS: CRC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motus Cleansing System (MCS) (Experimental): The MCS enables colon cleansing during standard colonoscopy using a standard colonoscope. The cleansing device, which is attached to the tip of the colonoscope and is connected to an external workstation, generates fluid jets within the colon thus dissolving the feces into small parts. The fecal matter & fluids are drained through the evacuation pipe of the cleansing device into a collecting reservoir.
  Interventions: Device: Motus Cleansing System

INTERVENTIONS:
Device: Motus Cleansing System

SUMMARY:
The Motus GI Colon Cleansing device is intended to facilitate intra-procedural cleaning of a poorly prepared colon by irrigating the colon and evacuating the irrigation fluid and feces.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the performance of the Motus cleansing system used in conjunction with screening, diagnostic or surveillance colonoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects being considered for diagnostic, screening or surveillance colonoscopy
2. Subjects in the age range of 18-75 years inclusive
3. Subjects with Body Mass Index (BMI) within the range of 18.5-35 inclusive
4. Subject has signed the informed consent

Exclusion Criteria:

1. Subjects with known Inflammatory Bowel Disease
2. Subjects with known diverticulitis disease or with prior incomplete colonoscopy due to diverticular disease
3. Subjects with known or detected (during colonoscopy) bowel obstruction
4. History of prior surgery to colon and/or rectum
5. ASA≥IV
6. Renal insufficiency (Creatinine ≥ 1.5mg /dL) (based on medical history)
7. Abnormal Liver enzymes (ALT/AST ≥ 2 times upper limits of normal) (based on medical history)
8. Subjects taking anticoagulants drugs (excluding aspirin) and dual anti-platelet therapy
9. Pregnancy (as stated by patient) or breast feeding
10. Subjects with altered mental status/inability to provide informed consent
11. Patients who have participated in another interventional clinical study in the last 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2017-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, PHD, Principal Investigator — HaEmek Medical Center, Afula Israel
Locations (1):
- HaEemek Medical Center, Afula, IL, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients recruited between Feb 2016 to Dec 2016 at "Emek Medical Center", Afula Israel.
Period: Overall Study
Arm/Group | Motus Cleansing System (MCS)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: patients indicate for colonoscopy procedure for screening, surveillance or/ and diagnosis.
Groups:
- Motus Cleansing System (MCS): The MCS enables colon cleansing during standard colonoscopy using a standard colonoscope. The cleansing device, which is attached to the tip of the colonoscope and is connected to an external workstation, generates fluid jets within the colon thus dissolving the feces into small parts. The fecal matter & fluids are drained through the evacuation pipe of the cleansing device into a collecting reservoir.
  Motus Cleansing System
Arm/Group | Motus Cleansing System (MCS)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 46.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Boston Bowel Preparation Scale( BBPS) >1 in All Colon Segments After the Use of MCS
Description: The rating of the cleansing quality was evaluated by using the Boston Bowel Preparation Scale (BBPS), Segment score of 0-3 given to each of the 3 segments of the colon (Left side, Transverse and right side):
  Score 0- Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  Score 1- A portion of the mucosa of the colon segment is seen, but other areas of the colon segment are not seen well due to staining, residual stool, and/or opaque liquid.
  Score 2- A minor amount of residual staining, small fragments of stool, and/or opaque liquid are visible, but the mucosa of the colon segment are seen well.
  Score 3-The entire mucosa of the colon segment is seen well with no residual staining, small fragments of stool, or opaque liquid.
  subject consider as having adequate cleaning if BBPS>1 in all colon segments
Time Frame: Within 24 hours- During the colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Motus Cleansing System (MCS)
Number analyzed (Participants) | 9
Participants | 9
Statistical Analysis 1: Comparison: Motus Cleansing System (MCS); patients had partial bowel preparation to mimic poor bowel cleansing before the colonoscopy procedure at baseline, MCS was used during the procedure to clean the colon; Test type: Other — Pilot study- no sample size was calculated; number of subjects with adequate cleansi = 100, 95% CI 2-sided [66 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Motus Cleansing System (MCS)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less